CLINICAL TRIAL: NCT03051672
Title: A Phase II Study Of Pembrolizumab In Combination With Palliative Radiotherapy For Metastatic Hormone Receptor Positive Breast Cancer
Brief Title: Phase II PEMBROLIZUMAB + PALLIATIVE RADIOTHERAPY IN BC
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Based on two-stage design, the study ended at stage 1 with no evidence of promise based on pre-specified decision rule.
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Sara Tolaney, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 16-588
Record Dates: First submitted 2017-02-08; First posted 2017-02-14 (Actual); Results first posted 2021-04-27 (Actual); Last update posted 2021-04-27 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Breast Cancer
Keywords: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Pembrolizumab With Radiation (Experimental): pembrolizumab : 200 mg intravenously 2 to 7 days prior to radiotherapy (RT) and on day 1 of repeating 21-day cycles. Treatment up to 35 cycles.
  Palliative radiation: a total dose of 20 Gy in 5 fractions
  Interventions: Drug: Pembrolizumab; Radiation: Palliative radiotherapy

INTERVENTIONS:
Drug: Pembrolizumab — Pembrolizumab (formerly MK-3475) is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD1 and its ligands, PD-L1 and PD-L2.
  Other Names: Keytruda
Radiation: Palliative radiotherapy — Palliative radiotherapy aims to shrink cancer, slow down its growth or control symptoms.

SUMMARY:
This research study is studying radiation therapy in combination with an immunotherapy as a possible treatment for metastatic hormone receptor (HR) positive, HER2-negative breast cancer.

The interventions involved in this study are:

* Palliative Radiotherapy
* Pembrolizumab

DETAILED DESCRIPTION:
This research study is a Phase II clinical trial. Phase II clinical trials test the safety and effectiveness of an investigational intervention to learn whether the intervention works in treating a specific disease. "Investigational" means that the intervention is being studied.

In this research study, the investigators are evaluating the safety and effectiveness of palliative radiotherapy ("radiation therapy") in combination with pembrolizumab in HR-positive, HER2-negative breast cancer. This study is designed to test how well radiation therapy in combination with pembrolizumab treats this type of cancer.

The FDA has approved radiation therapy as a treatment option for this type of breast cancer.

The FDA (the U.S. Food and Drug Administration) has not approved pembrolizumab for this specific disease but it has been approved in the United Sates for other types of cancer.

Pembrolizumab is a drug that may treat cancer by working with the immune system. The immune system is the body's natural defense against disease. The immune system sends types of cells called "T cells" throughout the body to detect and fight infections and diseases, including cancer. For some types of cancer, the T cells do not work as they should and are prevented from attacking the tumors. Pembrolizumab is thought to work by blocking a protein in the T cells called PD-1 ("programmed death 1"), which then allows these cells and other parts of the immune system to attack tumors.

The combination of pembrolizumab and radiation therapy is investigational. The study drug and radiation therapy, when given separately, work in different waysto help stop the cancer cells from growing and spreading. However, it is not known if giving the study drug and radiation therapy at the same time will have a better anti-cancer effect than giving each treatment on its own.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have histologically or cytologically confirmed invasive breast cancer, with metastatic disease. Participants without pathologic or cytologic confirmation of metastatic disease should have unequivocal evidence of metastasis from physical examination or radiologic evaluation.
* Invasive disease must have been tested for ER, PR and HER2. Participants must have hormone-receptor positive, HER2-negative breast cancer defined as:

  * ER>1% or PR>1%
  * HER2-negative per ASCO CAP guidelines, 2013 [Wolff et al., 2013]
* Participant must be a candidate for palliative radiation treatment to at least one bone, lymph node, or soft tissue lesion. Radiation of visceral lesions (such as lung or hepatic lesions) is not permitted.
* Participant must have measurable disease outside the field of radiation as defined by RECIST 1.1.
* If tumor is accessible and outside the field of radiation, the participant must be willing to undergo a research biopsy at baseline and after 2 cycles of pembrolizumab. Participants for whom newly-obtained samples cannot be provided (e.g. inaccessible or safety concern) must be willing to submit an archival specimen.
* Prior systemic therapy:

  * Participant must be at least 14 days from the last dose of prior chemotherapy, endocrine therapy, biological agents (including small molecule targeted therapy) or any investigational drug product with adequate recovery of toxicity to baseline, or grade 1(with the exception of alopecia and hot flashes) at the time of registration.
  * There is no limit to the number of prior lines of therapy, including endocrine or cytotoxic agents. Systemic treatment naive patients for metastatic disease are also eligible.
  * Participants may initiate or continue bisphosphonate therapy on study.
  * Continuation of ovarian suppression is allowed.
* Prior radiation therapy:

  * Patients must be at least 3 months from prior radiation therapy
  * Re-irradiation of the same field is not allowed
* Concurrent administration of other cancer specific therapy during the course of this study is not allowed.
* The subject is ≥18 years old
* ECOG performance status ≤1 (See Appendix A for details)
* Participants must have normal organ and marrow function as defined below:

  * absolute neutrophil count ≥1,500/mcL
  * platelets ≥100,000/mcL
  * hemoglobin ≥ 8 g/dl
  * total bilirubin ≤1.5 × institutional upper limit of normal (ULN)
  * AST(SGOT)/ALT(SGPT) ≤2.5 × institutional ULN or ≤ 5 × institutional ULN for participants with documented liver metastases
  * creatinine ≤1.5 ×within normal institutional ULN (or 2.0 x ULN in patients with documented Gilbert's Syndrome) OR creatinine clearance ≥60 mL/min/1.73 m2 for participants with creatinine levels above institutional ULN.
  * International normalized ratio (INR) or Prothrombin Time (PT) <1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
  * Activated Partial Thromboplastin Time (aPTT) <1.5 times the upper limit of normal unless subject is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended use of anticoagulants.
* Female subjects of childbearing potential must have a negative pregnancy test at screening
* Female and male subjects of childbearing potential must agree to use an adequate method of contraception as outlined in section 5.4.1. Contraception is required starting with the first dose of study medication through 120 days after the last dose of study medication Note: Abstinence is acceptable if this is the usual lifestyle and preferred contraception for the subject.
* Resolution of all chemotherapy-related or radiation-related toxicities to Grade 1 severity or lower, except for stable sensory neuropathy (≤ Grade 2) and alopecia.
* The subject is capable of understanding and complying with the protocol and has signed the informed consent document

Exclusion Criteria:

* Participants who are receiving any other investigational agents.
* Previous treatment with any anti-PD-1, PD-L1, or PD-L2 agent.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pembrolizumab.
* Known brain metastases that are untreated, symptomatic, or require therapy to control symptoms. Participants with previously diagnosed brain metastases are eligible if they have:

  * completed treatment (whole brain radiotherapy, radiosurgery, or a combination) at least 3 months prior to trial therapy initiation,
  * are neurologically stable, and
  * have recovered from effects of radiotherapy or surgery. Any corticosteroid use for brain metastases must have been discontinued without the subsequent appearance of symptoms for ≥2 weeks before prior to registration.
* Radiologic or clinical evidence of Spinal Cord Compression.
* Spinal Instability Neoplastic Score ≥ 7 unless lesion reviewed by a neurosurgical service and considered stable.
* Participants with bone lesions requiring surgical fixation to provide mechanical stability are ineligible. Participants with previously fixed lesions are allowed.
* The participant has an uncontrolled intercurrent illness, including, but not limited to uncontrolled hypertension, unstable angina pectoris, uncontrolled cardiac arrhythmia, congestive heart failure-New York Heart Association Class III or IV, active ischemic heart disease, myocardial infarction within the previous six months, uncontrolled diabetes mellitus, gastric or duodenal ulceration diagnosed within the previous 6 months, severe malnutrition or psychiatric illness/social situations that would limit compliance with study requirements.
* Clinically significant electrocardiogram (ECG) abnormality, including a marked baseline prolonged QT/QTc ([QT interval/corrected QT interval], eg, a repeated demonstration of a QTc interval >500 ms).
* Participant has a medical condition that requires chronic systemic steroid therapy or on any other form of immunosuppressive medication. For example, patients with autoimmune disease that requires systemic steroids or immunosuppression agents should be excluded. Replacement therapy (eg., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc.) is not considered a form of systemic treatment.
* Has history of (non-infectious) pneumonitis that required steroids or current pneumonitis.
* Has a history of interstitial lung disease.
* The participant is known to be positive for the human immunodeficiency virus (HIV), HepBsAg, or HCV RNA. HIV-positive participants on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Pembrolizumab.
* Individuals with a history of different malignancy are ineligible except for the following circumstances. Individuals with a history of other malignancies are eligible if they have been disease-free for at least 3 years or are deemed by the investigator to be at low risk for recurrence of that malignancy.
* Has received a live vaccine within 30 days of planned start of study therapy.
* The participant is pregnant or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2017-05-22 (Actual); Primary Completion 2018-09-04 (Actual); Study Completion 2019-01-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sara Tolaney, MD, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Barroso-Sousa R, Krop IE, Trippa L, Tan-Wasielewski Z, Li T, Osmani W, Andrews C, Dillon D, Richardson ET 3rd, Pastorello RG, Winer EP, Mittendorf EA, Bellon JR, Schoenfeld JD, Tolaney SM. A Phase II Study of Pembrolizumab in Combination With Palliative Radiotherapy for Hormone Receptor-positive Metastatic Breast Cancer. Clin Breast Cancer. 2020 Jun;20(3):238-245. doi: 10.1016/j.clbc.2020.01.012. Epub 2020 Jan 30. PMID 32113750

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients enrolled from May, 2017 to July, 2018.
Groups:
- Pembrolizumab With Radiation: Pembrolizumab will be administered intravenously prior to radiation pembrolizumab : 200 mg intravenously 2 to 7 days prior to radiotherapy (RT) and on day 1 of repeating 21-day cycles.
  Palliative radiation: a total dose of 20 Gy in 5 fractions
Period: Overall Study
Arm/Group | Pembrolizumab With Radiation
Started | 8
Began Treatment | 8
Completed | 8
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Pembrolizumab With Radiation: * Pembrolizumab will be administered intravenously prior to radiation
  * Pembrolizumab will be administered every 21 days
  * Palliative radiotherapy will be given for 5 treatments
Arm/Group | Pembrolizumab With Radiation
Number analyzed (Participants) | 8
Age, Continuous [Median (Full Range); unit: years] | 59 [37 to 68]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 8
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 8
  More than one race | 0
  Unknown or Not Reported | 0
ECOG Performance Status at Baseline [Count of Participants; unit: Participants] — Eastern Cooperative Oncology Group performance status, scaled 0 - 4.
  Participants
    0 - Normal activity | 2
    1 - Symptoms, but ambulatory | 6
    2 - In bed <50% of the time | 0
Site of Disease [Number; unit: case]
  CNS | 0
  Lung or pleural effusion | 2
  Liver | 5
  Bone | 8
  Breast or chest wall | 1
  Lymph nodes | 1
  Soft tissue | 0
  Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: The objective response rate (ORR) was defined as the proportion of participants achieving complete response (CR) or partial response (PR) outside the field of radiation based on RECIST 1.1 criteria on treatment. Per RECIST 1.1 for target lesions: CR is complete disappearance of all target lesions and PR is at least a 30% decrease in the sum of longest diameter (LD) of target lesions, taking as reference baseline sum LD. PR or better overall response assumes at a minimum incomplete response/stable disease (SD) for the evaluation of non-target lesions and absence of new lesions. Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: Tumor measurements are repeated every 6 weeks for the first 24 weeks and then every 9 weeks thereafter. Treatment continued until disease progression or unacceptable toxicity. Treatment duration was 1 cycle. Response was evaluated up to 3 months.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Pembrolizumab With Radiation
Number analyzed (Participants) | 8
percentage of participants | 0 [0 to 31.25]
Statistical Analysis 1: Comparison: Pembrolizumab With Radiation; The study uses a Simon 2-stage design. In stage 1, if >/=1 of 8 achieved OR then continue to stage 2 (enroll 19 more). If >/= 3 of 27 respond, the regimen would be considered promising. The null ORR<= 3% and alternative ORR>/=20%. With this design, the probability of stopping the trial early is 58% if the true ORR is 3%. This design at 80% power to declare the combination effective, while controlling for less than 5% 1-sided type I error under the null hypothesis; Test type: Superiority; The study terminated at stage 1 and no p-value was estimated; The study terminated at stage 1 and no p-value was estimated

2. Secondary Outcome: Incidence of Grade 4 Treatment-Related Toxicity
Description: All grade 4 adverse events (AE) with treatment attribution of possibly, probably or definite based on CTCAEv3 as reported on case report forms were counted. Incidence is the number of patients experiencing at least one treatment-related grade 4 AE of any type during the time of observation.
Time Frame: Tumor measurements are repeated every 6 weeks for the first 24 weeks and then every 9 weeks thereafter. Treatment continued until disease progression or unacceptable toxicity. Response was evaluated up to 3 months.
Measure: Number; unit: participants
Arm/Group | Pembrolizumab With Radiation
Number analyzed (Participants) | 8
participants | 0

3. Secondary Outcome: Median Progression-free Survival (PFS)
Description: Progression-free survival based on the Kaplan-Meier method is defined as the duration of time from study entry to documented disease progression (PD) or death. Per RECIST 1.1 criteria: progressive disease (PD) is at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions. PD for the evaluation of non-target lesions is the appearance of one or more new lesions and/or unequivocal progression of non-target lesions.
Time Frame: Tumor measurements are repeated every 6 weeks for the first 24 weeks and then every 9 weeks thereafter. Treatment continued until disease progression or unacceptable toxicity. The maximum follow-up time is 3 months.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Pembrolizumab With Radiation
Number analyzed (Participants) | 8
months | 1.4 [0.4 to 2.1]

4. Secondary Outcome: Median Overall Survival (OS)
Description: OS based on the Kaplan-Meier method is defined as the time from study entry to death or censored at date last known alive.
Time Frame: Tumor measurements are repeated every 6 weeks for the first 24 weeks and then every 9 weeks thereafter. Treatment continued until disease progression or unacceptable toxicity. The maximum follow-up time is 13 months.
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Pembrolizumab With Radiation: pembrolizumab : 200 mg intravenously 2 to 7 days prior to radiotherapy (RT) and on day 1 of repeating 21-day cycles.
  Palliative radiation: a total dose of 20 Gy in 5 fractions
  Pembrolizumab: Pembrolizumab (formerly MK-3475) is a potent and highly selective humanized monoclonal antibody (mAb) of the IgG4/kappa isotype designed to directly block the interaction between PD1 and its ligands, PD-L1 and PD-L2.
  Palliative radiotherapy: Palliative radiotherapy aims to shrink cancer, slow down its growth or control symptoms.
Arm/Group | Pembrolizumab With Radiation
Number analyzed (Participants) | 8
Months | 2.9 [0.9 to 3.6]

ADVERSE EVENTS:
Time Frame: AE data collected every cycle (21 days) from time of the first dose of study treatment, through the study and until removal from study or death, whichever occurs first. AEs were observed up to 3 months.
Description: Serious AEs (SAE) were defined as events with treatment-attribution of possibly, probably or definitely and grade 3 or higher. All remaining AEs are classified as Other AEs (OAE) including grade 3 or higher events with treatment-attribution of unlikely and unrelated plus all grade 1 and 2 events. Maximum grade toxicity by type was then calculated within SAE and OAE datasets. No further data is available to specify classification of other beyond the general term.
Arm/Group | Pembrolizumab With Radiation
All-Cause Mortality (participants affected / at risk) | 0/8
Serious Adverse Events (participants affected / at risk) | 0/8
Other Adverse Events (participants affected / at risk) | 7/8
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pembrolizumab With Radiation (N=8)
Vertigo (Ear and labyrinth disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 1
Metabolism and nutrition disorders - Other (Metabolism and nutrition disorders) | 1
Anemia (Blood and lymphatic system disorders) | 2
Hyperthyroidism (Endocrine disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Eye disorders - Other, specify (Eye disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 2
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Fatigue (General disorders) | 5
Flu like symptoms (General disorders) | 1
Pain (General disorders) | 1
Upper respiratory infection (Infections and infestations) | 1
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 4
Platelet count decreased (Investigations) | 1
Anorexia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 2
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bone pain (Musculoskeletal and connective tissue disorders) | 2
Osteoporosis (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 2
Anxiety (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-04-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03051672/Prot_SAP_000.pdf